CLINICAL TRIAL: NCT00781040
Title: Neutropenic Fever, Inflammatory Markers and Sepsis in Haematological Patients
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Sari Hamalainen, MD, PhD, Kuopio University Hospital
Other Study IDs: KUH5101409
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Sepsis
Keywords: Severe sepsis in neutropenic haematological patients
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neutropenic patients: Adult AML and ASCT patients with neutropenic fever.
  Interventions: Other: Severe sepsis vs. non-severe sepsis

INTERVENTIONS:
Other: Severe sepsis vs. non-severe sepsis — To compare these two groups
  Other Names: Severe sepsis vs. non-severe sepsis adult AML patients; Severe sepsis vs. non-severe sepsis adult ASCT patients

SUMMARY:
The aim of this study is to find out whether inflammation markers including cardiac markers have predictive value in evaluation of pathogenesis of sepsis in neutropenic haematological patients.

DETAILED DESCRIPTION:
Adult AML and ASCT patients with neutropenic fever. Observation of possible progress to severe sepsis or septic shock. Blood sample collection on days 0-3 (from the beginning of neutropenic fever).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis: acute myeloid leukaemia
* age under 70 years
* neutropenic fever

Exclusion Criteria:

* age above 70 years
* no neutropenic fever

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neutropenic patients in haematology ward having neutropenic fever with or without severe sepsis
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2006-12; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
This study evaluates epidemiology, microbiology and outcome of neutropenic fever and severe sepsis in haematological patients with special reference to the kinetics of inflammatory markers. | Within neutropenic period after treatment
  This study evaluated epidemiology, microbiology and outcome of neutropenic fever and severe sepsis in haematological patients with special reference to the kinetics of specific inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Esa Jantunen, M.D, PhD, Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanska M, Koivula I, Hamalainen S, Pulkki K, Nousiainen T, Jantunen E, Juutilainen A. High pentraxin 3 level predicts septic shock and bacteremia at the onset of febrile neutropenia after intensive chemotherapy of hematologic patients. Haematologica. 2011 Sep;96(9):1385-9. doi: 10.3324/haematol.2011.044925. PMID 21880642